CLINICAL TRIAL: NCT00390559
Title: Effects of Transdermal Nicotine on Tobacco Withdrawal and the Effects of Smoking-related Stimuli in Men and Women
Brief Title: Examining the Effect of the Nicotine Patch in Male and Female Smokers - 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NIDA-11082-3; R01DA011082 (NIH); R01-11082-3 DPMC
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Drug Addiction; Smoking Cessation
Keywords: Nicotine Replacement Therapy; Tobacco Smoking; Smoking stimuli; Gender
MeSH Terms: conditions — Substance-Related Disorders; Smoking Cessation; Tobacco Smoking; Coitus | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ActiveP/ActiveC (Experimental): 21 mg patch/Nicotine-containing cigarette
  Interventions: Drug: nicotine transdermal system; Other: Nicotine containing cigarette
- PlaceboP/ActiveC (Experimental): 0 mg patch/nicotine-containing cigarette
  Interventions: Drug: Nicotine transdermal system; Other: Nicotine containing cigarette
- Active P/PlaceboC (Experimental): 21 mg patch/no nicotine cigarette
  Interventions: Drug: nicotine transdermal system; Other: Placebo cigarette
- PlaceboP/PlaceboC (Experimental): 0 mg patch/no nicotine cigarette
  Interventions: Drug: Nicotine transdermal system; Other: Placebo cigarette

INTERVENTIONS:
Drug: nicotine transdermal system — 21 mg nicotine transdermal system
  Other Names: Nicoderm CQ
  Arms: Active P/PlaceboC; ActiveP/ActiveC
Drug: Nicotine transdermal system — Placebo nicotine patch
  Arms: PlaceboP/ActiveC; PlaceboP/PlaceboC
Other: Nicotine containing cigarette — Nicotine containing cigarette
  Arms: ActiveP/ActiveC; PlaceboP/ActiveC
Other: Placebo cigarette — Non nicotine containing cigarette
  Arms: Active P/PlaceboC; PlaceboP/PlaceboC

SUMMARY:
Treatment studies have demonstrated that current smoking cessation techniques are less effective for women. The purpose of this study is to determine the role that gender plays in the effectiveness of nicotine replacement therapy. In addition, the purpose of this study is to determine whether men and women differ in their response to smoking-related stimuli (e.g., taste or smell of a lit cigarette). Conclusions drawn from this study may help to improve cessation interventions for all smokers, particularly women.

DETAILED DESCRIPTION:
Currently,about 70 percent of smokers who try to quit by using smoking cessation treatments are unsuccessful. Treatment studies have demonstrated that current smoking cessation techniques are less effective for women. There is no clear explanation for this difference, but it may involve a differential response to nicotine replacement treatments (NRTs) and/or smoking-related stimuli. For women, NRT may be less effective at suppressing withdrawal or blunting the effects of smoking during a quit attempt. Women may also be more sensitive to smoking-related stimuli, suc has the taste, sight, or smell of cigarette smoke. Tailoring treatments to the separate needs of smoker subgroups , such as men and women, my produce better cessation outcomes. The purpose of this study is to assess whether men and women differ in the their response to NRT (i.e., transdermal nicotine) and smoking-related stimuli.

Participants in this double-blind, dose-comparison study will complete separate sessions in random order.

Each session will last approximately 6.5 hours and will correspond to a transdermal patch dose (0 or 21mg) and cigarette type (denicotinized and nicotinized). Objectively verified cigarette abstinence will be required before each session. Sessions will occur at least 48 hours apart to avoid carryover. At the beginning of each session a patch will be placed on the participant's back and at 4, 5, and 6 hours after patch application the participant will smoke a cigarette (all identifying marking on the cigarette will be covered for blinding purposes). Physiological, subjective, cognitive, and smoking behavior outcomes will be collected during study visits.

ELIGIBILITY:
Inclusion Criteria include, but are not limited to:

18-50 years of age Smokes 15 cigarettes/day for at least 2 years Healthy (as determined by a brief study physical with medical doctor) Displays understanding of cognitive tasks.

Exclusion Criteria include, but are not limited to:

History of chronic health problems or psychiatric conditions History of cardiovascular disease, low or high blood pressure, seizures, head injuries requiring hospital care, peptic ulcer, or diabetes Pregnancy (tested by urinalysis) Scores greater than 17 on the Beck Depression Inventory Lack of a high school degree or GED

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Eissenberg, PhD, Principal Investigator — Virginia Commonwealth University Department of Psychology, Institute for Drug and Alcohol Studies
Locations (1):
- Virginia Commonwealth University - Clinical Behavioral Pharmacology Laboratory, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment via media advertisement and flyer. Recruitment began 9/14/2005 and ended 1/30/2008.
Pre-assignment Details: Enrolled (i.e., consented) participants were excluded if they failed to meet safety criteria (e.g., blood pressure) measured after the informed consent was given.
Groups:
- All Participants: In this study, overnight abstinent smokers completed four, double-blind laboratory sessions corresponding to a 2x2 design where transdermal nicotine dose (TN, 0 or 21 mg) was crossed with type of cigarette (nicotine-containing [NIC] or not [DENIC]). Cigarettes were smoked 4 hours after TN administration.
Period: Overall Study
Arm/Group | All Participants
Started | 124
Received PlaceboP/Active C | 93
ActiveP/ActiveC | 87
PlaceboP/PlaceboC | 93
ActiveP/PlaceboC | 90
Completed | 80
Not Completed | 44

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 124
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 82

OUTCOME MEASURES:

1. Primary Outcome: Subjective Effects
Description: The full scale name is the "Urge to smoke" visual analog scale (VAS). It measures self-reported "urge to smoke". As with any VAS a word or phrase (in this case, "Urge to Smoke" is centered over a horizontal line anchored on the left by "not at all" and on the right by "extremely." In this study, participants used a mouse to produce a vertical mark on the horizontal line, and the score was the distance of the mark from the left anchor expressed as a percentage of total line length. Thus, the minimum was 0 ("not at all") and the maximum score was 100 ("extremely").
Time Frame: 6 hours
Population: Those who completed all four "arms" of the crossover study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ActiveP/ActiveC | PlaceboP/ActiveC | Active P/PlaceboC | PlaceboP/PlaceboC
Number analyzed (Participants) | 80 | 80 | 80 | 80
units on a scale | 18.8 (24.7) | 23.1 (24.5) | 25.6 (28.8) | 24.2 (25.8)

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | ActiveP/ActiveC | PlaceboP/ActiveC | Active P/PlaceboC | PlaceboP/PlaceboC
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No